CLINICAL TRIAL: NCT05134571
Title: A Phase 4, Single-arm, Open-label Safety and Efficacy Study of Aldurazyme® (Laronidase) as Enzyme Replacement Therapy in Participants With Mucopolysaccharidosis I (MPS I) in China
Brief Title: China Post-marketing Surveillance (PMS) Study of Aldurazyme®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS16578; U1111-1260-3947 (Registry Identifier: ICTRP)
Record Dates: First submitted 2021-10-21; First posted 2021-11-26 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Mucopolysaccharidosis I
Keywords: clinical trial; enzyme replacement therapy; mucopolysaccharidosis I; laronidase
MeSH Terms: conditions — Mucopolysaccharidosis I | interventions — Iduronidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Aldurazyme (laronidase) (Experimental): Aldurazyme (laronidase) treatment at approved dose and regimen, administered every week as an IV infusion
  Interventions: Drug: Laronidase

INTERVENTIONS:
Drug: Laronidase — Solution for injection; Intravenous

SUMMARY:
This is a single treatment arm study that is open-label to be conducted in Chinese participants with MPS I.

Trial Objectives are to evaluate the safety and tolerability of Aldurazyme in Chinese MPS I participants, and to evaluate the efficacy of Aldurazyme on the percent change of urinary glycosaminoglycans (uGAGs) from baseline to Week 26. The study will also evaluate the effect on uGAG level and liver volume (hepatomegaly) after 26 weeks, with Aldurazyme treatment in Chinese MPS I participants.

Treatment duration will include: 2 weeks of screening, 26 weeks of treatment and 1 week of follow-up period. During the treatment period, weekly visits are designed to accommodate weekly administration of Aldurazyme (laronidase).

DETAILED DESCRIPTION:
Study duration for each participant will be a total of 29 weeks which will include 2 weeks of screening, 26 weeks of treatment period and 1 week of follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Chinese participants have a documented diagnosis of MPS I confirmed by measurable clinical signs and symptoms of MPS I and fibroblast or leukocyte IDUA (iduronidase) activity <10% of normal.
* Participants have to be able to stand independently and walk a minimum of 5 meters in 6 minutes.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

  * Is not a woman of childbearing potential (WOCBP).
  * OR
  * Is a WOCBP and agrees to use an acceptable contraceptive method during the intervention period and at a minimum until 7 days after the last dose of study intervention.
  * A WOCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) within the screening period before the first dose of study intervention.
  * If a urine test cannot be confirmed as negative (eg, an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
  * Contraceptive/barrier method is not applicable for male participants.

Exclusion Criteria:

* Prior tracheostomy or bone marrow transplantation or hematopoietic stem cell transplantation.
* Have a plan to undergo bone marrow transplantation or hematopoietic stem cell transplantation within half a year after enrollment.
* Received an investigational drug, or device, other than Aldurazyme, within 30 days prior to study enrollment.
* Received an investigational gene therapy.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Participants with adverse events (AEs) | Baseline to Week 27
  Incidence of AEs, serious adverse events (SAEs) and adverse events of special interest (AESIs) including infusion associated reactions (IARs) during the treatment emergent (TE) period
The incidence of Potentially clinically significant abnormality (PCSA) analyses for clinical laboratory, vital signs, and ECG parameters during the TE period | Baseline to Week 27
The percent change of uGAGs | Baseline to Week 26

SECONDARY OUTCOMES:
The percent change of uGAGs | Baseline to Week 2, Week 4, Week 8, Week 12 and Week 20
The absolute change of uGAGs | Baseline to Week 2, Week 4, Week 8, Week 12, Week 20 and Week 26
The percent change of liver volume (Abdominal B type ultrasound examination) | Baseline to Week 26

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (5):
- China (5):
  - Investigational Site Number :1560003, Beijing
  - Investigational Site Number :1560002, Beijing
  - Investigational Site Number :1560004, Guangzhou
  - Investigational Site Number :1560006, Hangzhou
  - Investigational Site Number :1560001, Wuhan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Liang Y, Yang YL, Zou CC, Liu L, Jiao Y, Wang Y, Liu X, Luo XP. Safety and efficacy of laronidase in Chinese patients with mucopolysaccharidosis type I: a phase IV, single-arm, open-label, multicenter study. Orphanet J Rare Dis. 2025 Oct 29;20(1):547. doi: 10.1186/s13023-025-04056-w. PMID 41163043
- See also: LPS16578 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25282&tenant=MT_SNY_9011